CLINICAL TRIAL: NCT02850549
Title: Implementation of a Neck Pain Classification System: A Preliminary Analysis
Brief Title: Preliminary Neck Classification Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Ambrose University (Other)
Responsible Party: Principal Investigator, Kevin Farrell, Principal Investigator, St. Ambrose University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StAmbroseU2
Record Dates: First submitted 2016-07-26; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Neck Pain
Keywords: neck pain; cervical; classification; outcomes; physical therapy
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- physical therapy (Other): Physical Therapy intervention provided by therapists in phase one without training in following a neck classification system and in phase two after being trained to follow a neck pain classification system.
  Interventions: Other: Procedure: physical therapy and Neck Pain Classification

INTERVENTIONS:
Other: Procedure: physical therapy and Neck Pain Classification — Physical therapists treated patients in phase one as they usually do and in phase two were trained to follow a neck classification and matched intervention system.

SUMMARY:
The purpose of this study was to assess if pain and function in patients with neck pain is less when physical therapists use a classification system.

DETAILED DESCRIPTION:
The purpose of this study was to prospectively assess pain and function scores in patients with neck pain, with therapists specifically trained to implement a treatment based classification and matched interventions system. This study consisted of two phases to determine whether implementing a classification changed patient outcomes. In phase one, baseline data was obtained while physical therapists continued with their current neck pain evaluation and intervention approaches. The second phase involved educating the therapists in the neck classification system with the matched interventions. Pain and function outcomes were analyzed for 2 phases. The overall goal was to prospectively determine if the implementation of this classification system with matched interventions could enhance patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Licensed physical therapists
* Treat patients with neck pain on a regular basis

Exclusion Criteria:

* Do not utilize interventions included in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating (NPR) | up to 107 days
  NPR was measured on initial evaluation and at the time the patient was discharged from care which varied for each patient (ranged from 3 to 107 days).
Neck Disability Index (NDI) | up to 107 days
  NDI was measured on initial evaluation and at the time the patient was discharged from care which varied for each patient (ranged from 3 to 107 days).

SECONDARY OUTCOMES:
Number of Visits | Measured from initial evaluation to time of discharge from care; up to 107 days.
Duration of Care | Number of days of care, measured from initial evaluation to time of discharge from care; up to 107 days.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Farrell, Principal Investigator — St. Ambrose University
Locations (7):
- United States (7):
  - Genesis Physical Therapy - King Plaza, Moline, Illinois
  - Genesis Physical Therapy - Illini, Silvis, Illinois
  - Genesis Physical Therapy - Maplecrest, Bettendorf, Iowa
  - Genesis Physical Therapy - Lombard, Davenport, Iowa
  - Genesis Physical Therapy - 53rd St, Davenport, Iowa
  - Genesis Physical Therapy - Valley Fair, Davenport, Iowa
  - Genesis Physical Therapy - Le Claire, Le Claire, Iowa

IPD SHARING:
Plan to Share IPD: No